CLINICAL TRIAL: NCT06731634
Title: Prevalence of De Quervain' S Tenosynovit's Syndrome Among Egyptian Medical Students with Smart Phone Addiction
Brief Title: De Quervain Syndrome Among Medical Students with Smart Phone Addiction
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basil Aly Zaky Aly Amer, Physiotherapist at the egyption ministry of health, Cairo University
Other Study IDs: 012/005462
Record Dates: First submitted 2024-12-03; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: De Quervain Tenosynovitis; Smartphone Addiction
Keywords: De quervain tenosynovitis; Egyptian medical students; Cairo University; Smartphone addiction; Prevelance
MeSH Terms: conditions — De Quervain Disease; Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- One group will be assigned: The group will include people with smartphone addiction, who will receive a Finkelstein test for both dominant and non dominant hand, then the both hands grip and bench strength will be tested.
  Interventions: Device: Hand grip strength dynamometer, pinch strength dynamometer; Diagnostic Test: Finkelstein test

INTERVENTIONS:
Device: Hand grip strength dynamometer, pinch strength dynamometer — Both devices will be used to assign the strength of grip and pinch for both dominant and non dominant hands by using jamar hydraulic hand grip strength dynamometer and Jamar hydraulic pinch strength dynamometer
Diagnostic Test: Finkelstein test — Finkelstein test which is used to diagnose the de quervain tenosynovitis and it will be used to assist the people with smartphone addiction

SUMMARY:
To investigate the prevelance of the de quervain tenosynovitis among the Egyptian medical students with smartphone addiction

DETAILED DESCRIPTION:
Addictive participants will be assigned and enrolled in the study according to there addiction score on smartphone addiction scale.

Participants will receive a Finkelstein test for both dominant and non dominant hand for the de quervain tenosynovitis.

Then the strentgh of both hand grip and pinch grip for both hands will be tested using hand grip strength dynamometer and pinch strentgh dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic students with normal healthy state
* Any student in all the academic years with age 18-25
* Addictive smart phone users with score over 31 for male and 33 for female students in smart phone addiction scale.
* Who own or use mobile.
* Both genders: male and female
* Willing to participate.
* Egyptian students

Exclusion Criteria:

* Those who don't have mobile phone.
* Any previous injury or trauma or surgery and a history of rheumatoid arthritis, osteoarthritis, and deformities and changes in the shape of the finger joints.
* Those who are not willing to participate.
* Non-Egyptian students.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be recruited from the medical collages of Cairo University in Egypt
Sampling Method: Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dominant hand grip strength and Non-Dominant hand grip strength by the using of jamar hydraulic grip strength dynamometer | 1 Day
Dominant hand pinch strength and non-dominant hand pinch strength by the using of jamar hydraulic pinch strength dynamometer | 1 Day

SECONDARY OUTCOMES:
The degree of pain during the finkelstein test by the using of visual analoug scale | 1 Day
  The visual analoug scale (vas) will be used to identify the degree of pain that the participant felt during the finkelstein test the scale values are from 0mm to 100mm 0mm means he didn't feel any pain which is good, 100mm means he felt the morst pain which is bad

IPD SHARING:
Plan to Share IPD: Undecided